CLINICAL TRIAL: NCT06925399
Title: Dynamic Changes of Innate Immune Cells in Pregnant Women With Autoimmune Thyroid Disease
Brief Title: Changes in Natural Immunity in Pregnant Women With Autoimmune Thyroid Disease
Acronym: CIPAT
Status: Not yet recruiting | Type: Observational
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Tatjana Bogović Crnčić, Associate professor, MD, PhD, Head of the Department of Nuclear Medicine at Faculty of Medicine, University of Rijeka
Other Study IDs: uniri-iskusni-biomed-23-61
Record Dates: First submitted 2025-03-19; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy; Autoimmune Thyroid Disease
Keywords: Pregnancy; Autoimmune thyroid disease; Innate immunity; NKT cells; Monocytes; Neutrophils

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women referred for thyroid examination due to suspected thyroid disease: Adult pregnant women referred to the Clinical Department of Nuclear Medicine and the Department of Endocrinology, Diabetes and Metabolic Diseases of the Clinic of Internal Medicine of the Clinical Hospital Center Rijeka for thyroid examination due to suspected or known AITD and who have signed an informed consent form will participate in the study. The following data is collected and analyzed from pregnant women who are included in the examination on the basis of a signed consent form: Age, number of pregnancies, number of abortions, pregnancy outcome (abortion, premature birth, timely birth, delayed birth). The pregnant women included in the study will be tested three times, i.e. in the first, second and third trimester of pregnancy. Depending on the results of the hormone status and the thyroid autoantibody titre, the pregnant women will be divided into two groups: (1) normal pregnancy and (2) pregnant women with autoimmune thyroid disease.

SUMMARY:
Autoimmune thyroid disease (AITD) is the most common endocrine disorder in women of reproductive age, including during pregnancy. It encompasses two clinical conditions: autoimmune hyperthyroidism and hypothyroidism. Pregnancy significantly affects thyroid function regulation, while thyroid dysfunction can influence fertility, pregnancy progression, and the postpartum health. Although the role of acquired immunity in AITD is well understood, recent research increasingly emphasizes innate immunity. Key cells involved in innate immunity include neutrophils, monocytes, and NKT cells. However, limited data exist on their role during pregnancy, especially in women with AITD.

This study aims to investigate the dynamic changes in neutrophils, monocytes and NKT cells during pregnancy and compare findings between women with normal pregnancies and those with AITD.

The study will analyze the frequency and activation status of these innate immune cells in peripheral blood samples collected during the first, second, and third trimesters. In addition, concentrations of thyrotropin, thyroid hormones, thyroglobulin, and thyroid autoantibodies, will be measured. A thyroid ultrasound will also be performed.

DETAILED DESCRIPTION:
Autoimmune thyroid disease (AITD) affects approximately 2-17% of women of reproductive age, and represents the most common endocrine disorder in pregnancy. It includes autoimmune hyperthyroidism and hypothyroidism. Pregnancy has a significant impact on the regulation of thyroid function, and thyroid dysfunction may contribute to adverse pregnancy outcomes and neonatal complications.

Early detection of thyroid dysfunction during pregnancy is critical for optimal maternal-fetal health. While acquired immunity is a recognized contributor to the development of AITD, increasing attention has been given to the role of innate immunity. Innate immune mechanisms are essential for early immune response initiation and maintaining maternal tolerance toward the fetus, which represents a semi-allogeneic entity. This tolerogenic state is regulated both systemically and locally at the maternal-fetal interface.

The most relevant innate immune cells include neutrophils, monocytes/macrophages, and natural killer T (NKT) cells. Neutrophils participate in immune defense through cytotoxicity, phagocytosis, and cytokine secretion. Their numbers increase during pregnancy, and they play a role in implantation and placental development. Monocytes and decidual macrophages contribute to immune tolerance and placental remodeling. NKT cells, which bridge innate and adaptive immunity, perform immunoregulatory functions and have been observed in increased proportions in the decidua compared to peripheral blood. However, limited data are available regarding their role in pregnancy with thyroid autoimmunity.

The hypothesis of this study is that the numbers of neutrophils, monocytes and NKT cells and activation state of monocytes and NKT cells change during normal pregnancy and in pregnancy affected by AITD. The primary objective is to analyze differences in the frequency and activation marker expression of these immune cells between the two groups.

Peripheral blood mononuclear cells will be isolated, labeled, and analyzed using flow cytometry.

Expression of HLA-DR on monocytes and CD69 and CD25 on NKT cells will be quantified. In parallel, thyroid function parameters will be measured, including thyrotropin (TSH), free thyroxine (FT4), free triiodothyronine (FT3), thyroglobulin (Tg), and thyroid autoantibodies (TPOAb, TgAb, antiTSHR).

Pregnant women will be enrolled prospectively and will undergo blood sampling in each trimester. Ultrasound evaluation of the thyroid gland will be conducted to aid in diagnosis and classification. Participants will be categorized into groups based on thyroid hormone status and autoantibody titers: (1) normal pregnancy and (2) pregnancy with AITD.

The expected enrollment is 80 pregnant women (40 per group). All analyses will be conducted according to standardized laboratory and immunophenotyping protocols.

Statistical analysis will include group comparisons using t-tests or ANOVA for parametric data and Mann-Whitney or Kruskal-Wallis tests for non-parametric data. Correlation analyses will be conducted using Pearson or Spearman coefficients. A p-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria: adult healthy pregnant women and pregnant women with autoimmune thyroid disease

* with a single pregnancy
* older than 18 years
* who have signed the informed consent form

Exclusion Criteria:

* pregnant women who refuse to give informed consent
* pregnant women under the age of 18
* pregnant women with malignant diseases
* pregnant women with thyrotoxicosis or hypothyroidism of a non-autoimmune nature and previous thyroidectomy or ablative therapy with iodine-131
* pregnant women with an acute or chronic disease that is not an autoimmune thyroid disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only adult pregnant women are eligible for the study
Study Population: The planned prospective observational study will include pregnant women referred by primary care clinics in Rijeka and Primorsko-goranska County to the Clinical Department of Nuclear Medicine and the Department of Endocrinology, Diabetes and Metabolic Diseases of the Clinic of Internal Medicine of the Clinical Hospital Center Rijeka for thyroid examination and who have signed an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of Neutrophils in Peripheral Blood | Within 24 months from enrollment; analysis over a 12-month period.
  Frequency of neutrophils will be measured by differential blood count. Unit of Measure: Percent (%)
Frequency of Monocytes in Peripheral Blood | Within 24 months from enrollment; analysis over a 12-month period.
  Monocyte frequency will be measured by flow cytometry and expressed as percentage of monocytes among CD45⁺ leukocytes.
  Unit of Measure: Percent (%)
Frequency of NKT Cells in Peripheral Blood | Within 24 months from enrollment; analysis over a 12-month period.
  NKT cell frequency will be measured by flow cytometry and expressed as percentage of NKT cells within CD3⁺ T lymphocytes.
  Unit of Measure: Percent (%)

SECONDARY OUTCOMES:
Expression of HLA-DR on Monocytes | Within 24 months from enrollment.
  HLA-DR expression on CD14⁺ monocytes will be measured using flow cytometry and expressed as percentage of HLA-DR⁺ monocytes.
  Unit of Measure: Percent (%)
Expression of CD25 on NKT Cells | Within 24 months from enrollment.
  CD25 expression on CD3⁺CD56⁺ NKT cells will be measured using flow cytometry and expressed as percentage of CD25⁺ cells.
  Unit of Measure: Percent (%)
Expression of CD69 on NKT Cells | Time Frame: Within 24 months from enrollment.
  CD69 expression on CD3⁺CD56⁺ NKT cells will be measured using flow cytometry and expressed as percentage of CD69⁺ cells.
  Unit of Measure: Percent (%)
Serum Concentration of TSH | Measured at each trimester; analysis completed within 12 months of final collection.
  TSH concentration will be measured using a chemiluminescent immunoassay (CLIA). Unit of Measure: mU/L
Serum Concentration of Free T4 | Measured at each trimester; analysis completed within 12 months.
  Unit of Measure: pmol/L
Serum Concentration of Free T3 | Measured at each trimester; analysis completed within 12 months.
  Unit of Measure: pmol/L
Serum Concentration of Thyroglobulin (Tg) | Measured at each trimester; analysis completed within 12 months.
  Unit of Measure: ng/mL
Serum Concentration of TPOAb | Measured at each trimester; analysis completed within 12 months.
  Unit of Measure: IU/mL
Serum Concentration of TgAb | Measured at each trimester; analysis completed within 12 months.
  Unit of Measure: IU/mL
Serum Concentration of antiTSHR | Measured at each trimester; analysis completed within 12 months.
  Unit of Measure: IU/L

OTHER OUTCOMES:
Correlation Between Immune Cell Frequencies and Thyroid Biomarkers | Within 24 months from enrollment.
  Correlation between neutrophil, monocyte, and NKT cell frequencies and thyroid hormone/antibody levels.
  Unit of Measure: Correlation coefficient (r)
Correlation Between Activation Marker Expression and Thyroid Biomarkers | Within 24 months from enrollment.
  Correlation between expression of HLA-DR, CD25, and CD69 and thyroid hormone/antibody levels.
  Unit of Measure: Correlation coefficient (r)
Gestational Age at Delivery | Time Frame: At delivery
  Unit of Measure: Weeks
Birth Weight | Time Frame: At delivery
  Unit of Measure: Grams
Preterm Birth Occurrence | At delivery
  Unit of Measure: Yes/No
Correlation Between Immune Cell Parameters and Pregnancy Outcomes | Within 24 months from enrollment.
  Correlation between immune cell parameters and pregnancy outcomes such as gestational age, preterm birth, and birth weight.
  Unit of Measure: Correlation coefficient (r)

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Bogović Crnčić, Principal Investigator — Faculty of Medicine University of Rijeka
Locations (1):
- Faculty of Medicine University of Rijeka, Clinical Hospital Center Rijeka, Rijeka, Primorsko-goranska County, Croatia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available upon request from Tatjana Bogović Crnčić
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: The principal investigator and collaborators involved in the research will have access to the IPD and supporting information.
  Working versions of the data will be stored during the project on the principal investigator's computer, the project collaborator's laptop, and an external drive to which both the collaborators and the principal investigator will have access.
  The final version of the data will be made available by the principal investigator through the repository of the Faculty of Medicine in Rijeka, established in the national Dabar system, where publications and other project documents will be stored.